CLINICAL TRIAL: NCT03856710
Title: A Double-blinded Randomised Controlled Trial Comparing the Clinical and Cost Effectiveness of Self-fixating Versus Stapled Mesh in the Laparoscopic Management of Inguinal Hernia
Brief Title: Self Fixating Versus Stapled Mesh for Laparoscopic Inguinal Hernia Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Doncaster And Bassetlaw Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0874/2017/CTN
Record Dates: First submitted 2019-01-27; First posted 2019-02-27 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Inguinal Hernia
Keywords: Inguinal hernia; Groin hernia; Laparoscopy; Mesh
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Intervention Model Description: This is a double blinded randomised controlled trial of ProGripTM self-gripping mesh versus standard 'lightweight' (large pore) polypropylene mesh fixed with SecurestrapTM an absorbable strap fixation device in the laparoscopic treatment of inguinal hernias. Sample size is 47 patients per group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be unaware of the type of mesh received as the randomisation process will be carried out intraoperatively when the patient is under general anaesthesia. Subsequently, over the follow-up period every possible effort will be made to continue the blinding process in order to minimise any bias in patient reported outcomes. Similarly outcome assessors would be blinded as well.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Self-gripping Mesh), (Active Comparator): The initial laparoscopic approach will be the same for both groups until the process of selection and placement of the mesh , which would be decided by randomization by sealed envelope. This group will receive self-gripping mesh
  Interventions: Device: self-gripping mesh
- Group 2 (Stapled Mesh) (Active Comparator): The initial laparoscopic approach will be the same for both groups until the process of selection and placement of the mesh , which would be decided by randomization by sealed envelope. This group will receive stapled mesh
  Interventions: Device: Stapled mesh

INTERVENTIONS:
Device: self-gripping mesh — The initial laparoscopic approach will be the same for both groups until the process of selection and placement of the mesh (ProGripTM self-gripping mesh versus standard 'lightweight' (large pore) polypropylene mesh fixed with SecurestrapTM) which would be decided by randomization by sealed envelope into one of the 2 intervention groups: Group 1 (Self-gripping Mesh), Group 2 (Stapled Mesh).
  Arms: Group 1 (Self-gripping Mesh),
Device: Stapled mesh — The initial laparoscopic approach will be the same for both groups until the process of selection and placement of the mesh (ProGripTM self-gripping mesh versus standard 'lightweight' (large pore) polypropylene mesh fixed with SecurestrapTM) which would be decided by randomization by sealed envelope into one of the 2 intervention groups: Group 1 (Self-gripping Mesh), Group 2 (Stapled Mesh).
  Arms: Group 2 (Stapled Mesh)

SUMMARY:
Inguinal (groin) hernias are common and occur when an internal part of the body pushes through a weakness in the surrounding tissue wall of the groin. They are more likely to occur in men and affect people's quality of life by causing pain that is worse after any strenuous activity. If untreated they can cause serious problems such as strangulation when too much bowel comes through the weakness and becomes squeezed with the risk of losing blood supply requiring emergency surgery. To prevent such complications, elective surgery for symptomatic inguinal hernias is undertaken either in the conventional open method which involves a cut in the groin, or the keyhole surgery, when the surgery is undertaken via three small incisions in the abdomen (instead of a single, larger groin incision), a thin tube containing a light source and a camera (laparoscope) is inserted through one of these incisions, so the surgeon can see inside the abdomen. Special surgical instruments are inserted through the other incisions, so the surgeon can pull or push the hernia back into place and a piece of mesh is then stapled or glued to secure it to the weakened area in the abdomen wall. Securing the mesh with staple has been associated with increased post-operative pain and analgesia requirement; whereas not doing so has been thought to increase the chances of recurrence- more so in large sized weakness. A newer mesh appears to offer benefit over conventional meshes as it grips the tissues around the weakness without requiring staples or glue to fix it in place, and has shown to cause lesser post-operative pain and recurrence.

This study is going to compare the newer self-gripping mesh with the conventional mesh requiring fixation to see which is best for patients undergoing keyhole repair to fix inguinal hernias.

DETAILED DESCRIPTION:
Design: Double Blinded Randomised Controlled Trial This is a multicentre randomised controlled trial in the setting of two district general teaching hospitals serving an aggregate population of over 750 000. There are already established general surgical clinics and operating sessions available for and including study patients. Both units undertake conventional open and laparoscopic treatments for inguinal hernias on a regular basis in keeping with the national average numbers.

Methodology; Patients with symptomatic unilateral or bilateral inguinal hernias diagnosed clinically &/or radiologically will be identified at general surgical clinics and the primary investigator, will arrange the following;

* Assess inclusion / exclusion criteria for participation in study
* Informed written consent for participation in the study
* Baseline clinical severity and quality of life analysis using:

  * Euroqol (EQ5D)
  * Core Outcome Measures Index adapted for patients with hernia (COMI-hernia)
* Informed written consent for intervention (the patient will be blinded as to the intervention group) Subjects; Patients will be identified during attendance to our general surgical clinics. Patients will be clearly informed that participation in the study is entirely voluntary and that refusal to participate will in no way disadvantage them.

Intervention (within 3 months of randomization);

* Re-assess inclusion / exclusion criteria
* Ensure informed written consent for surgery / participation in the study
* Intervention; The initial laparoscopic approach will be the same for both groups until the process of selection and placement of the mesh (ProGripTM self-gripping mesh versus standard 'lightweight' (large pore) polypropylene mesh fixed with SecurestrapTM) which would be decided by randomization by sealed envelope into one of the 2 intervention groups: Group 1 (Self-gripping Mesh), Group 2 (Stapled Mesh). The surgeon will have a choice of Transabdominal Preperitoneal (TAPP) or Total Extraperitoneal (TEP) to perform the laparoscopic inguinal hernia repair. Both TAPP and TEP are standard laparoscopic techniques used for treatment of inguinal hernias both within the National Health Service (NHS) and across the world.

Postoperative Care Since most laparoscopic inguinal hernia repairs are performed as day cases, patients may be discharged on the same day of surgery after recovery with simple analgesia. Diet can be resumed immediately and the convalescent period is expected to be 1-2 days with routine activities expected to resume at 2 weeks.

Blinding precautions:

Patients will be unaware of the type of mesh received as the randomisation process will be carried out intraoperatively when the patient is under general anaesthesia. Subsequently, over the follow-up period every possible effort will be made to continue the blinding process in order to minimise any bias in patient reported outcomes.

Perioperative outcome measures

* Time taken for procedure
* Admission / 30-day readmission rates
* Procedure-specific complications
* Direct (marginal) costs Post-operative assessments Performed at 1 week, 6 weeks, 3 months and 12 months (by Surgical Registrar blinded to the intervention received by the patient). 1 Week and 3 month follow-up will be over telephone (with a view to review patient in the Hospital, should any concerns be expressed or elicited from the patient); 6 weeks and 12 month follow-up will be face-to-face in an out-patient clinic setting.

At each assessment the following will be analysed:

1. Pain - recorded prospectively in a diary by the patient independently. Recorded daily for the first week on an un-marked 100mm long scale, from absolutely no pain to the worst imaginable pain
2. Analgesia requirements - recorded daily for the first week in a diary by the patient independently
3. Extent of ecchymosis, seroma/haematoma - The registrar will assess for any signs of ecchymosis, seroma or haematoma and measure the magnitude of surface area(s) affected at 6 weeks.
4. Time to return to work and normal activities - reported by the patient. (Post-op all patients will be advised to mobilise and return to normal activities as soon as they feel able)
5. Procedure-specific complications;
6. Clinical efficacy and effectiveness; using

   * Euroqol (EQ5D)
   * Core Outcome Measures Index adapted for patients with hernia (COMI-hernia)
   * Patient satisfaction rating scales
7. Cost effectiveness and cost benefit; using

   * Direct costs
   * Indirect costs
   * Willingness to pay data

Quality of life and economic analysis;

* Generic Euroqol (EQ5D) instrument
* Core Outcome Measures Index adapted for patients with hernia (COMI-hernia) The combination of these generic EQ5D and disease specific COMI-hernia tools are thus sensitive to assess & compare both multidimensional and cost-effectiveness outcomes in patients undergoing surgical treatment for inguinal hernia repair.
* Procedure-specific complications
* Patient satisfaction rating scale
* Cost effectiveness analysis; will be analysed in terms of

  * Cost / symptom-free patient
  * Cost / QALY (Quality-Adjusted Life Years) calculated from the EQ5D and COMI-hernia indices Direct hospital costs will be collected prospectively with the help of the hospital finance department; whilst indirect patient cost data (income loss, domestic support etc.) will be assessed and calculated at interview at 3 and 12 months. Direct & indirect costs will provide total costs for use in the cost/QALY calculations.
* Cost benefit analysis; outcomes, expressed as monetary units assessed by direct willingness to pay (WTP) questioning, at 3 and 12 months will be used for cost benefit analysis e.g. cost / £ willing to pay and cost / percent of weekly income willing to pay.

Data collection and analysis Data will be collected and entered onto a specifically designed Microsoft Access database Data distribution will be studied and analysed appropriately. Intergroup analysis will be performed using Mann-Whitney U test and intragroup analysis will be performed using the Friedman test across time points and Wilcoxon's ranked sum test between two time points. Regression techniques and multivariate analysis will then be utilised for a more thorough interrogation of the data.

For the economic analysis, the incremental cost per QALY of the intervention will be assessed. This follows the example of National Institute of Clinical Excellence (NICE) who use a threshold of £20 000 to £30 000 per QALY gained. However, cost-effectiveness analysis is conducted under conditions of uncertainty. Cost effectiveness acceptability curves (CEACs) will be generated to demonstrate the uncertainty around the decision. Given the data available within the model, the CEAC will plot the probability of one strategy being more cost-effective than the others for a range of threshold values of an additional QALY.

Interim Analysis:

An interim analysis will be carried out after recruitment of 25 patients per group. The goal of this analysis is to evaluate recruitment rates, adverse events and serious adverse events if any, as well as the overall viability and conduct of the trial.

The reported rates of moderate to severe chronic groin pain affecting QoL after elective hernia repair ranges between 0 to 36%8-11. The variation is also attributed to the inconsistencies in the definition of chronic pain. Investigators have taken the chronic pain rates from one of the larger reported series (Garg et al 200937) to calculate the sample size as their rates may be similar to the predicted chronic pain rates when fixing moderate to large sized defects with permanent fixation devices. The sample size of 47 per group (allowing for a dropout rate of 15%) will therefore be a pragmatic number to achieve recruitment, follow-up and completion of the trial within the anticipated time period. However the sample size derived from the meta-analysis (Sajid et al 201338) will be considered for a future multi-centre trial that is planned by investigators' group based on the outcomes from this pilot study.

Ethical issues;

* All patients will be given adequate time to read the patient information sheet
* No undue pressure will be exerted on any individual to participate in the study
* The patient consent form will be signed by the patient and the researcher, only when both are happy that the patient has understood the information sheet and is willing to give informed written consent to participate in the study, and that the patient understands that it is their right to withdraw from the trial at any time without prejudice to their future treatment.

Project milestones Based upon the average number of patients seen in general surgical clinics with symptomatic inguinal hernias requiring surgical intervention, we envision recruitment taking 6-8 months across both sites.

Taking an average waiting time of 3 months from clinic appointment to date of operation, most patients in the trial should have their planned intervention by 9-12 months from start of recruitment.

Most of the key outcomes will be collected within 6 weeks post procedure. The most important outcomes of chronic pain and early recurrence will be evaluated at 3, 12 month follow-up post procedure, hence taking between 18-24 months for completion of trial.

The effect sizes used for sample size calculation were conservative and the true required sample may be lower. An interim analysis will be performed after recruitment of 25 patients per group. This data will help to guide the requirement for further recruitment and establish if intergroup differences are larger than expected. It may be possible to curtail recruitment with a lower sample size.

Risk Profile It is not likely that there should be any reason to stop this trial prematurely, as the interventions in question are currently in regular clinical practice both in the NHS and worldwide without any added risks reported by the manufacturers or in the scientific literature.

Intervention; Both treatment techniques of laparoscopic fixation of mesh with stapling device and use of self-gripping mesh not requiring fixation are used already for treatment of inguinal hernias, both within the NHS and across the world. They have been shown to be safe and effective, with no more increase in complications. Treatment related risks will be covered by NHS indemnity.

Complications are classed as:

Non-specific: Acute post-operative pain, infection, haematoma, recurrence, port site hernia.

Specific complications: Chronic post-operative pain, shrinkage; dislocation; migration; erosion of mesh All procedures will be planned and performed by Consultant Surgeons skilled and experienced in the performance of laparoscopic inguinal hernia mesh repair. Complications and adverse events will be reported to the Principal Investigator and each incidence individually investigated. Any concerns over outcomes will be discussed with all of the co-investigators and clinicians involved in the trial. Any safety concerns will result in suspension of the trial pending further investigation.

Trial Process; All of the trial outcomes are non-invasive and offer no significant risk to patients; in fact the enhanced follow-up will allow closer monitoring of patients for procedure or product related complications.

The participants will have given their informed consent, prior to taking part in this study. All participant details will be number coded and kept securely. Participants are unlikely to be identified from digital images, which will be numbered to ensure anonymity and archived securely.

The overall aim is to observe and compare outcomes in patients undergoing standardised, established treatment protocols currently in wide utilisation, with no deviation from standard practice. As such investigators do not envisage patients being placed at undue risk.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Demonstrated to have primary or recurrent unilateral or bilateral inguinal hernia
* Both patient and surgeon occupy a position of equipoise over the relative merits of either intervention
* Ability to give informed written consent

Exclusion Criteria:

* Non-elective acute presentation with inguinal hernia and its complications
* Inability to give informed written consent
* Groin symptoms which on clinical examination and radiological investigations fail to demonstrate any evidence of inguinal hernia.
* Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2017-09-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Chronic pain rates Hernia recurrence rates | 12 months
  Pain persisting beyond 3 months post inguinal hernia surgery
Hernia recurrence rates | 12 months
  Clinical or radiological evidence of inguinal hernia at any time point

SECONDARY OUTCOMES:
Technical success | 1 day
  Both techniques will be compared for conversion from laparoscopic procedure to open.
Operative time | 1 day
  Both techniques will be compared for time taken to complete surgery (in minutes)
Analgesia requirement | 1 week
  Both techniques will be compared for analgesic consumption
Perioperative complications including injury to organs, bleeding | 1 day
  Both techniques will be compared for any perioperative complications.
Return to work and routine activities | 12 months
  Both techniques will be compared for time taken to return to work and routine activities( in days).
Quality-of-life improvement | 12 months
  Both techniques will be compared for improvement in quality of life using specified questionnaires
Cost effectiveness of the two techniques by assessing incremental cost per QALY of the intervention | 12 months
  Both techniques will be compared for cost effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Srinivasan Balchandra, MS, MD, FRCS, Principal Investigator — Doncaster and Bassetlaw Teaching Hospitals NHS Foundation trust
Locations (1):
- Doncaster and Bassetlaw Teaching Hospitals Nhs Foundation Trust, Doncaster, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The data will be utilised by the parent research team to make comparisons of the two techniques as listed in the protocol and results presented at scientific conferences and shared in the scientific literature. However sharing individual patient data has not been decided and in the future may be considered subject to data protection and confidentiality policies.
Supporting Information: Study Protocol
Time Frame: 6 months after the Trial completion and will be available for 2 years
Access Criteria: The study results will be shared with other researchers once completed. All listed and relevant participant Data, access criteria, statistics and clinical study report will be shared.